CLINICAL TRIAL: NCT03891901
Title: IMPACT-TB (Imatinib Mesylate Per Oral as a Clinical Therapeutic for TB): A Phase II Clinical Trial of the Safety, Pharmacokinetics and Hematologic Effects of Imatinib on Myelopoiesis in Adults When Given With and Without Isoniazid and Rifabutin
Brief Title: A Clinical Trial of the Safety, Pharmacokinetics and Hematologic Effects of Imatinib on Myelopoiesis in Adults When Given With and Without Isoniazid and Rifabutin
Acronym: IMPACT-TB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Emory University (Other); University of Pennsylvania (Other); Aurum Institute (Other); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Aim 1; 38518 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-08

CONDITIONS: Tuberculosis
Keywords: Imatinib; Rifabutin; Isoniazid
MeSH Terms: conditions — Tuberculosis | interventions — Imatinib Mesylate; Isoniazid; Rifabutin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid (Experimental): Participants will receive 50 mg imatinib for 14 days, followed by 14 days of imatinib together with rifabutin and isoniazid.
  Interventions: Drug: Imatinib; Drug: Isoniazid; Drug: Rifabutin
- Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid (Experimental): Participants will receive 100 mg imatinib for 14 days, followed by 14 days of imatinib together with rifabutin and isoniazid.
  Interventions: Drug: Imatinib; Drug: Isoniazid; Drug: Rifabutin
- Cohort 1c: Imatinib (200 mg) + Rifabutin + Isoniazid (Experimental): Participants will receive 200 mg imatinib for 14 days, followed by 14 days of imatinib together with rifabutin and isoniazid.
  Interventions: Drug: Imatinib; Drug: Isoniazid; Drug: Rifabutin
- Cohort 1d: Imatinib (400 mg) + Rifabutin + Isoniazid (Experimental): Participants will receive 400 mg imatinib for 14 days, followed by 14 days of imatinib together with rifabutin and isoniazid.
  Interventions: Drug: Imatinib; Drug: Isoniazid; Drug: Rifabutin
- Cohort 2a: Imatinib + Rifabutin + Isoniazid (Experimental): Participants will receive isoniazid and rifabutin for 14 days, followed by 14 days of combination isoniazid, rifabutin, and imatinib. Imatinib dose will be determined after analyzing data from Cohort 1.
  Interventions: Drug: Imatinib; Drug: Isoniazid; Drug: Rifabutin
- Cohort 2b: Imatinib + Rifabutin + Isoniazid (Experimental): Participants will receive isoniazid and rifabutin for 14 days, followed by 14 days of combination isoniazid, rifabutin, and imatinib. Imatinib dose will be determined after analyzing data from Cohort 1.
  Interventions: Drug: Imatinib; Drug: Isoniazid; Drug: Rifabutin
- Imatinib (100 mg) (Experimental): Participants will receive 100 mg imatinib daily for 28 days.
  Interventions: Drug: Imatinib
- Imatinib (200 mg) (Experimental): Participants will receive 200 mg imatinib daily for 28 days.
  Interventions: Drug: Imatinib
- Imatinib (400 mg) (Experimental): Participants will receive 400 mg imatinib daily for 28 days.
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Tablets, administered orally
Drug: Isoniazid — 300 mg tablets, administered orally
  Arms: Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid; Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid; Cohort 1c: Imatinib (200 mg) + Rifabutin + Isoniazid; Cohort 1d: Imatinib (400 mg) + Rifabutin + Isoniazid; Cohort 2a: Imatinib + Rifabutin + Isoniazid; Cohort 2b: Imatinib + Rifabutin + Isoniazid
Drug: Rifabutin — 300 mg capsules, administered orally
  Arms: Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid; Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid; Cohort 1c: Imatinib (200 mg) + Rifabutin + Isoniazid; Cohort 1d: Imatinib (400 mg) + Rifabutin + Isoniazid; Cohort 2a: Imatinib + Rifabutin + Isoniazid; Cohort 2b: Imatinib + Rifabutin + Isoniazid

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics, and effects of imatinib on myelopoiesis in adults when given with and without isoniazid and rifabutin. The results of this trial will determine the imatinib dose to be studied in a subsequent Phase IIB treatment trial of imatinib as an adjunctive therapy with an antimicrobial regimen (rifabutin, pyrazinamide (PZA), isoniazid (INH) and ethambutol) for drug-sensitive TB.

DETAILED DESCRIPTION:
With existing anti-tubercular drug therapies, treatment of drug-susceptible TB takes at least 6 months and success rates for multi-drug resistant tuberculosis (MDR-TB) and extensively drug resistant TB (XDR-TB) are a dismal 50 and 20%, respectively, highlighting the urgent need for new TB drugs. The cancer drug imatinib limits mycobacterial infections in culture and animal models by reducing both entry into macrophages and augmenting phagolysosomal fusion (autophagy), which may facilitate antigen presentation and pathogen killing. Additionally, imatinib induces increases in myeloid cells (myelopoiesis), and an innate immune response to infection that mimics so-called "emergency hematopoiesis," a response that Mycobacterium tuberculosis (Mtb) appears to suppress. Importantly, these mechanisms can be induced in animal models by oral doses substantially lower than those used in people to combat cancer. The dose-dependence has important implications for TB clinical studies in humans, as it suggests that imatinib could improve TB treatment using doses that impart minimal, if any, toxicity.

This study will evaluate the safety, pharmacokinetics, and effects of imatinib on myelopoiesis in adults when given with and without isoniazid and rifabutin (antibiotics to treat mycobacterial infections).

Participants will be enrolled into one of two cohorts. In Cohort 1, participants will be enrolled in a dose-escalating fashion to receive one of four doses of imatinib alone for 14 days, followed by imatinib in combination with rifabutin and isoniazid for another 14 days.

In Cohort 2, participants will receive rifabutin and isoniazid for 14 days, followed by 14 days of rifabutin and isoniazid in combination with one of the two selected doses of imatinib. The exact doses of imatinib administered in Cohort 2 will be determined after analyzing data from Cohort 1.

After safety evaluations of participants enrolled into the first two dose levels of Cohort 1, the intervention of imatinib followed by imatinib in combination with rifabutin and isoniazid was discontinued. The study protocol was amended to evaluate the effects of imatinib alone, at 3 escalating doses.

Total study duration for participants will be 50 days, during which time participants will attend several study visits. Study visits may include a physical exam, electrocardiogram, blood and urine collection, and pharmacokinetic assessments.

ELIGIBILITY:
Inclusion Criteria:

* Adult age between 18 years and 55 years
* Body mass index (BMI) greater than 18.5 kg/m^2
* At least 8 years formal education, with appropriate reading and comprehension skills
* Able and willing to provide written informed consent
* Males must agree to using contraception during the study and for 2 weeks after the last dose of study drug.
* If a female participant is of reproductive potential, the participant (and her partner) must agree to use of one of the following combinations of birth control during the study and for 2 weeks after the last dose of study drug (or tubal ligation as a single method):

  * Use of a double-barrier method of contraception: condoms (male or female) and a diaphragm or cervical cap with spermicide;
  * Use of an intrauterine device (IUD) and a barrier method: condoms (male or female, with or without spermicide) or a diaphragm or cervical cap with spermicide;
  * For those in the imatinib only study arms: use of hormone-based contraceptives (pill, patch, implant, ring, or injectable) and a barrier method: condoms (male or female, with or without spermicide) or a diaphragm or cervical cap with spermicide (participants in study arms receiving isoniazid and rifabutin are not eligible if they are relying hormonal contraceptives other than an IUD)
  * Tubal ligation.
  * Women who are post-menopausal, defined as age greater than 45 and no menses for at least 1 year, or who have had a hysterectomy, are considered not of reproductive potential.

Exclusion Criteria:

* Current or imminent treatment for significant infection
* Pregnant or breastfeeding
* HIV positive status as determined by a U.S. Food and Drug Administration (FDA)-approved HIV assay
* Hepatitis B infection, as determined by an FDA-approved hepatitis B surface antigen assay
* Hepatitis C infection, as determined by an FDA-approved positive Hepatitis C antibody assay
* Known infection with Mycobacterium tuberculosis (MTB)
* History of allergy or hypersensitivity to imatinib, isoniazid or rifabutin.
* History of enrollment in other clinical trials with investigational agents within 8 weeks
* Cardiac arrhythmia requiring medication, or any clinically significant electrocardiogram (ECG) abnormality
* Exam consistent with congestive heart failure (e.g., edema)
* Random blood glucose greater than 140 mg/dL or history of unstable diabetes mellitus requiring hospitalization for hyper or hypoglycemia within the past year prior to start of screening
* Use of systemic corticosteroids within the past 28 days
* Any of the following readings from a complete blood count that fall outside the normal ranges as listed here:

  * White blood cell count: 3.4 10E3/microliter (mcL) - 11 10E3/mcL
  * Hemoglobin: Female- 11.1 - 16.7 gm/dL, Male- 12.5 - 16.5 gm/dL
  * Platelet count: 150-400 10E3/mcL
  * Absolute neutrophil count: Female- 0.91-5.53 10E3/mcL, Male- 0.67-6.41 10E3/mcL
  * Absolute lymphocyte count: Female- 0.65-3.05 10E3/mcL, Male- 0.72-3.29 10E3/mcL
* Any of the following chemistry panel and liver function test readings that fall outside the normal ranges as listed here:

  * Serum potassium: 3.5-5.4 mmol/L
  * Alkaline phosphatase (ALP): 34 - 104 unit/L
  * Alanine aminotransferase (ALT): 4 - 52 unit/L
  * Aspartate aminotransferase (AST): 13 - 39 unit/L
  * Total Bilirubin: 0.2 - 1.0 mg/dL
  * Creatinine: Female- 0.60-1.20 mg/dL, Male- 0.7-1.3mg/dL
* Cirrhosis of the liver, or any known active or chronic liver disease
* Current or past alcohol or elicit/recreational drug use, which in the expert judgment of the Investigator, will interfere with the participant's ability to comply with the protocol requirements.
* Any experimental medications for less than 8 weeks prior to screening or anticipated use during the trial
* Current (within 30 days prior to the first dose of study drug) or anticipated use of antimetabolites; alkylating agents; or other drugs or herbal preparations (including St. John's wort), known to affect activity of the CYP3A4 enzyme pathway
* Consumption of grapefruit, grapefruit juice, or grapefruit-related citrus fruits (e.g., pomelos) within 7 days before assessment for eligibility
* Unwilling to avoid grapefruit or grapefruit-related citrus fruits/pomelo during the course of the study
* Unwilling to avoid alcohol for the duration of the study
* Unwilling to abstain from taking acetaminophen-containing medications during the 28-day study drug dosing period, due to increased risk of liver toxicity
* History of major medical disorders including metabolic, endocrine, hypothyroid, hepatic, renal, hematologic, pulmonary, gastrointestinal, autoimmune or cardiovascular disorders
* Uncontrolled hypertension (persistent measurements at or above 150/100)
* Participants who are, in the opinion of the Investigator, unable to comply with the dosing schedule and protocol evaluations
* Diarrhea defined as 4 or more stools per day
* Active involvement (by the participant or the participant's partner) in In Vitro Fertilization or another assisted reproductive technology procedure
* Emory students currently enrolled in a course taught by the principal investigator (PI) or a Co-Investigator
* Emory employees currently working under supervision of the PI or a Co-Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edmund K. Waller, MD, PhD, FACP, Principal Investigator — Emory University School of Medicine, Winship Cancer Institute
Locations (1):
- Emory University DAIDS TB Non-Network CRS, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through the Winship Cancer Institute, Georgia Clinical & Translational Science Alliance (Georgia CTSA) Clinical Research Center, and Emory University Hospital in Atlanta, Georgia, USA. Participant enrollment began on October 27, 2020 and study visits were completed by August 30, 2022.
Pre-assignment Details: A total of 42 individuals were screened and 18 did not meet eligibility criteria or withdrew prior to the baseline assessment, resulting in 24 study participants initiating study activities.
Groups:
- Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid: Participants receiving 50 mg imatinib for 14 days, followed by 14 days of imatinib together with rifabutin and isoniazid.
  Imatinib: Tablets, administered orally
  Isoniazid: 300 mg tablets, administered orally
  Rifabutin: 300 mg capsules, administered orally
- Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid: Participants receiving 100 mg imatinib for 14 days, followed by 14 days of imatinib together with rifabutin and isoniazid.
  Imatinib: Tablets, administered orally
  Isoniazid: 300 mg tablets, administered orally
  Rifabutin: 300 mg capsules, administered orally
- Cohort 1c: Imatinib (200 mg) + Rifabutin + Isoniazid: Participants receiving 200 mg imatinib for 14 days, followed by 14 days of imatinib together with rifabutin and isoniazid.
  Imatinib: Tablets, administered orally
  Isoniazid: 300 mg tablets, administered orally
  Rifabutin: 300 mg capsules, administered orally
- Cohort 1d: Imatinib (400 mg) + Rifabutin + Isoniazid: Participants receiving 400 mg imatinib for 14 days, followed by 14 days of imatinib together with rifabutin and isoniazid.
  Imatinib: Tablets, administered orally
  Isoniazid: 300 mg tablets, administered orally
  Rifabutin: 300 mg capsules, administered orally
- Cohort 2a: Imatinib + Rifabutin + Isoniazid; Cohort 2b: Imatinib + Rifabutin + Isoniazid: Participants receiving isoniazid and rifabutin for 14 days, followed by 14 days of combination isoniazid, rifabutin, and imatinib. Imatinib dose will be determined after analyzing data from Cohort 1.
  Imatinib: Tablets, administered orally
  Isoniazid: 300 mg tablets, administered orally
  Rifabutin: 300 mg capsules, administered orally
- Imatinib (100 mg): Participants receiving 100 mg imatinib daily for 28 days.
  Imatinib: Tablets, administered orally
- Imatinib (200 mg): Participants receiving 200 mg imatinib daily for 28 days.
  Imatinib: Tablets, administered orally
- Imatinib (400 mg): Participants receiving 400 mg imatinib daily for 28 days.
  Imatinib: Tablets, administered orally
Period: Overall Study
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid | Cohort 1c: Imatinib (200 mg) + Rifabutin + Isoniazid | Cohort 1d: Imatinib (400 mg) + Rifabutin + Isoniazid | Cohort 2a: Imatinib + Rifabutin + Isoniazid | Cohort 2b: Imatinib + Rifabutin + Isoniazid | Imatinib (100 mg) | Imatinib (200 mg) | Imatinib (400 mg)
Started | 16 | 6 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Began Imatinib Plus Rifabutin and Isoniazid Portion of the Intervention (if Applicable) | 14 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 12 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not Completed | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Exposure to coronavirus disease 2019 (COVID-19) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Poor venous access | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid: Participants receiving 50 mg imatinib for 14 days, followed by 14 days of imatinib together with rifabutin and isoniazid.
- Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid: Participants receiving 100 mg imatinib for 14 days, followed by 14 days of imatinib together with rifabutin and isoniazid.
- Imatinib (100 mg): Participants receiving 100 mg imatinib daily for 28 days.
- Total: Total of all reporting groups
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid | Imatinib (100 mg) | Total
Number analyzed (Participants) | 16 | 6 | 2 | 24
Age, Customized [Count of Participants; unit: Participants]
  18-25 years | 7 | 3 | 0 | 10
  26-35 years | 7 | 1 | 1 | 9
  36-45 years | 2 | 0 | 0 | 2
  46-55 years | 0 | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 2 | 16
  Male | 5 | 3 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 15 | 5 | 2 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 0 | 7
  White | 8 | 4 | 2 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 6 | 2 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Myelomonocytic Cells in the Blood
Description: Immunologic effects of the study treatment are assessed by counting myelomonocytic cells in blood samples. An increase in myelomonocytic cells is used to determine the appropriate therapeutic dose of imatinib.
Time Frame: Days 1, 7, 14, 21, 28, 42
Population: The analysis population includes participants who completed the study.
Measure: Mean (Standard Deviation); unit: cells per microliter (µL)
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid | Imatinib (100 mg)
Number analyzed (Participants) | 12 | 2 | 2
cells per microliter (µL)
  Day 1 | 3197 (933) | 4340 (480) | 3390 (283)
  Day 7 | 3241 (1393) | 3680 (1414) | 3075 (64)
  Day 14 | 3418 (1640) | 3195 (1265) | 3195 (21)
  Day 21 | 3021 (1479) | 2560 (721) | 2785 (332)
  Day 28 | 2356 (1059) | 1140 (98) | 2480 (198)
  Day 42 | 3629 (1548) | 4425 (403) | 3255 (841)

2. Primary Outcome: Frequency of Grade 3 or 4 Adverse Events (AEs)
Description: The number of grade 3 or 4 adverse events occurring among study participants is presented here. Adverse events are graded using the FDA Guidance Document, "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials Guidance for Industry," September 2007, or other guidance, as applicable.
Time Frame: Measured through Day 50
Measure: Number; unit: Grade 3 or 4 adverse events
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid | Imatinib (100 mg)
Number analyzed (Participants) | 16 | 6 | 2
Grade 3 or 4 adverse events | 4 | 6 | 0

3. Primary Outcome: Frequency of Serious Adverse Events (SAEs)
Description: The number of serious adverse events occurring among study participants is presented here. Adverse events are graded using the FDA Guidance Document, "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials Guidance for Industry," September 2007, or other guidance, as applicable.
Time Frame: Measured through Day 50
Measure: Number; unit: serious adverse events
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid | Imatinib (100 mg)
Number analyzed (Participants) | 16 | 6 | 2
serious adverse events | 0 | 0 | 0

4. Secondary Outcome: White Blood Cell Count
Description: The normal range for white blood cell counts is between 4,000 and 11,000 cells per microliter. White blood cell counts increase during infections, autoimmune diseases and some types of cancer. Low white blood cell counts occur with immune system diseases and certain types of cancer.
Time Frame: Days 1, 7, 14, 21, 28, 42
Population: The analysis population includes participants who completed the study.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid | Imatinib (100 mg)
Number analyzed (Participants) | 12 | 2 | 2
cells/µL
  Day 1 | 5558 (1099) | 6300 (1272) | 5900 (566)
  Day 7 | 5391 (1222) | 5900 (1697) | 5500 (283)
  Day 14 | 5841 (1648) | 5150 (2192) | 5400 (1273)
  Day 21 | 4875 (1430) | 3650 (636) | 4750 (212)
  Day 28 | 4141 (1295) | 1600 (282) | 4800 (424)
  Day 42 | 5841 (1684) | 5800 (282) | 5300 (1414)

5. Secondary Outcome: Maximum Concentration (Cmax) of Imatinib
Description: Blood samples for pharmacokinetic (PK) analyses of imatinib were collected at 6 time points over approximately 24 hours. Samples collection occurred at hour 0 (pre-dose), and 0.5 hours, 2 hours, 4.0 hours, 8.0 hours, and 24 hours post-dose. PK samples were taken after 14 days of imatinib alone (all study arms) and after 14 days of imatinib with rifabutin and isoniazid (Cohorts 1a and 1b). The PK parameter Cmax is the highest concentration of imatinib in blood following dosing.
Time Frame: Day 14, Day 28
Population: The analysis population includes those who were participating in the study at the indicated time point. Participants in the Imatinib (100 mg) group, who received imatinib alone, had a single PK analysis.
Measure: Median (Inter-Quartile Range); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid | Imatinib (100 mg)
Number analyzed (Participants) | 14 | 4 | 2
micrograms per milliliter (mcg/mL)
  After 14 days of imatinib | 0.41 [0.27 to 0.69] | 0.69 [0.46 to 0.75] | 0.51 [0.48 to 0.54]
  After 14 days of imatinib plus rifabutin and isoniazid: number analyzed (Participants) | 12 | 2 | 0
  After 14 days of imatinib plus rifabutin and isoniazid | 0.71 [0.23 to 1.47] | 0.69 [0.66 to 0.72] |

6. Secondary Outcome: Half-life (T1/2) of Imatinib
Description: Blood samples for pharmacokinetic (PK) analyses of imatinib were collected at 6 time points over approximately 24 hours. Samples collection occurred at hour 0 (pre-dose), and 0.5 hours, 2 hours, 4.0 hours, 8.0 hours, and 24 hours post-dose. PK samples were taken after 14 days of imatinib alone (all study arms) and after 14 days of imatinib with rifabutin and isoniazid (Cohorts 1a and 1b). The PK parameter T1/2 is the time when imatinib in blood is half of the maximum concentration.
Time Frame: Day 14, Day 28
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid | Imatinib (100 mg)
Number analyzed (Participants) | 14 | 4 | 2
hours
  After 14 days of imatinib | 11.32 [8.20 to 16.47] | 15.01 [9.66 to 16.62] | 11.00 [10.62 to 11.37]
  After 14 days of imatinib plus rifabutin and isoniazid: number analyzed (Participants) | 12 | 2 | 0
  After 14 days of imatinib plus rifabutin and isoniazid | 9.91 [7.85 to 11.29] | 7.83 [7.01 to 8.65] |

7. Secondary Outcome: Area Under the Curve (AUC) for Imatinib
Description: Blood samples for pharmacokinetic (PK) analyses of imatinib were collected at 6 time points over approximately 24 hours. Samples collection occurred at hour 0 (pre-dose), and 0.5 hours, 2 hours, 4.0 hours, 8.0 hours, and 24 hours post-dose. PK samples were taken after 14 days of imatinib alone (all study arms) and after 14 days of imatinib with rifabutin and isoniazid (Cohorts 1a and 1b). The PK parameter AUC is the overall exposure to imatinib.
Time Frame: Day 14, Day 28
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: hour*mcg/mL
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid | Imatinib (100 mg)
Number analyzed (Participants) | 14 | 4 | 2
hour*mcg/mL
  After 14 days of imatinib | 4.76 [3.32 to 10.21] | 9.46 [6.42 to 12.53] | 5.80 [5.48 to 6.12]
  After 14 days of imatinib plus rifabutin and isoniazid: number analyzed (Participants) | 12 | 2 | 0
  After 14 days of imatinib plus rifabutin and isoniazid | 7.52 [2.69 to 16.59] | 7.49 [6.99 to 7.98] |

8. Secondary Outcome: Elimination Rate Constant (Ke) of Imatinib
Description: Blood samples for pharmacokinetic (PK) analyses of imatinib were collected at 6 time points over approximately 24 hours. Samples collection occurred at hour 0 (pre-dose), and 0.5 hours, 2 hours, 4.0 hours, 8.0 hours, and 24 hours post-dose. PK samples were taken after 14 days of imatinib alone (all study arms) and after 14 days of imatinib with rifabutin and isoniazid (Cohorts 1a and 1b). The elimination rate constant is the rate that imatinib is removed from the body.
Time Frame: Day 14, Day 28
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: 1/hour
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid | Imatinib (100 mg)
Number analyzed (Participants) | 14 | 4 | 2
1/hour
  After 14 days of imatinib | 0.06 [0.04 to 0.08] | 0.05 [0.04 to 0.07] | 0.06 [0.06 to 0.07]
  After 14 days of imatinib plus rifabutin and isoniazid: number analyzed (Participants) | 12 | 2 | 0
  After 14 days of imatinib plus rifabutin and isoniazid | 0.07 [0.06 to 0.09] | 0.09 [0.08 to 0.10] |

9. Secondary Outcome: Maximum Concentration (Cmax) of Isoniazid
Description: Blood samples for pharmacokinetic (PK) analyses of isoniazid were collected at 6 time points over approximately 24 hours. Samples collection occurred at hour 0 (pre-dose), and 0.5 hours, 2 hours, 4.0 hours, 8.0 hours, and 24 hours post-dose. PK samples were taken after 14 days of imatinib with rifabutin and isoniazid (Cohorts 1a and 1b). The PK parameter Cmax is the highest concentration of the drug in blood following dosing.
Time Frame: Day 28
Population: The analysis population includes those who completed the study. One participant was excluded from the Imatinib 50mg group due to unreliable PK parameters for isoniazid and rifabutin.
Measure: Median (Inter-Quartile Range); unit: mcg/mL
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid
Number analyzed (Participants) | 11 | 2
mcg/mL | 3.14 [1.88 to 4.97] | 3.66 [2.72 to 4.59]

10. Secondary Outcome: Half-life (T1/2) of Isoniazid
Description: Blood samples for pharmacokinetic (PK) analyses of isoniazid were collected at 6 time points over approximately 24 hours. Samples collection occurred at hour 0 (pre-dose), and 0.5 hours, 2 hours, 4.0 hours, 8.0 hours, and 24 hours post-dose. PK samples were taken after 14 days of imatinib with rifabutin and isoniazid (Cohorts 1a and 1b). The PK parameter T1/2 is the time when the drug in blood is half of the maximum concentration.
Time Frame: Day 28
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid
Number analyzed (Participants) | 11 | 2
hours | 1.59 [1.15 to 2.05] | 2.44 [2.33 to 2.55]

11. Secondary Outcome: Area Under the Curve (AUC) for Isoniazid
Description: Blood samples for pharmacokinetic (PK) analyses of isoniazid were collected at 6 time points over approximately 24 hours. Samples collection occurred at hour 0 (pre-dose), and 0.5 hours, 2 hours, 4.0 hours, 8.0 hours, and 24 hours post-dose. PK samples were taken after 14 days of imatinib with rifabutin and isoniazid (Cohorts 1a and 1b). The PK parameter AUC is the overall exposure to the drug.
Time Frame: Day 28
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: hour*mcg/mL
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid
Number analyzed (Participants) | 11 | 2
hour*mcg/mL | 9.79 [7.22 to 15.03] | 16.11 [12.74 to 19.48]

12. Secondary Outcome: Elimination Rate Constant (Ke) of Isoniazid
Description: Blood samples for pharmacokinetic (PK) analyses of isoniazid were collected at 6 time points over approximately 24 hours. Samples collection occurred at hour 0 (pre-dose), and 0.5 hours, 2 hours, 4.0 hours, 8.0 hours, and 24 hours post-dose. PK samples were taken after 14 days of imatinib with rifabutin and isoniazid (Cohorts 1a and 1b). The elimination rate constant is the rate that the drug is removed from the body.
Time Frame: Day 28
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: 1/hour
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid
Number analyzed (Participants) | 11 | 2
1/hour | 0.44 [0.34 to 0.60] | 0.28 [0.27 to 0.30]

13. Secondary Outcome: Maximum Concentration (Cmax) of Rifabutin
Description: Blood samples for pharmacokinetic (PK) analyses of rifabutin were collected at 6 time points over approximately 24 hours. Samples collection occurred at hour 0 (pre-dose), and 0.5 hours, 2 hours, 4.0 hours, 8.0 hours, and 24 hours post-dose. PK samples were taken after 14 days of imatinib with rifabutin and isoniazid (Cohorts 1a and 1b). The PK parameter Cmax is the highest concentration of the drug in blood following dosing.
Time Frame: Day 28
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: mcg/mL
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid
Number analyzed (Participants) | 11 | 2
mcg/mL | 0.37 [0.34 to 0.51] | 0.53 [0.47 to 0.60]

14. Secondary Outcome: Half-life (T1/2) of Rifabutin
Description: Blood samples for pharmacokinetic (PK) analyses of rifabutin were collected at 6 time points over approximately 24 hours. Samples collection occurred at hour 0 (pre-dose), and 0.5 hours, 2 hours, 4.0 hours, 8.0 hours, and 24 hours post-dose. PK samples were taken after 14 days of imatinib with rifabutin and isoniazid (Cohorts 1a and 1b). The PK parameter T1/2 is the time when the drug in blood is half of the maximum concentration.
Time Frame: Day 28
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid
Number analyzed (Participants) | 11 | 2
hours | 9.65 [7.38 to 10.91] | 8.14 [7.78 to 8.50]

15. Secondary Outcome: Area Under the Curve (AUC) for Rifabutin
Description: Blood samples for pharmacokinetic (PK) analyses of rifabutin were collected at 6 time points over approximately 24 hours. Samples collection occurred at hour 0 (pre-dose), and 0.5 hours, 2 hours, 4.0 hours, 8.0 hours, and 24 hours post-dose. PK samples were taken after 14 days of imatinib with rifabutin and isoniazid (Cohorts 1a and 1b). The PK parameter AUC is the overall exposure to the drug.
Time Frame: Day 28
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: hour*mcg/mL
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid
Number analyzed (Participants) | 11 | 2
hour*mcg/mL | 3.68 [2.89 to 5.20] | 5.11 [4.24 to 5.98]

16. Secondary Outcome: Elimination Rate Constant (Ke) of Rifabutin
Description: Blood samples for pharmacokinetic (PK) analyses of rifabutin were collected at 6 time points over approximately 24 hours. Samples collection occurred at hour 0 (pre-dose), and 0.5 hours, 2 hours, 4.0 hours, 8.0 hours, and 24 hours post-dose. PK samples were taken after 14 days of imatinib with rifabutin and isoniazid (Cohorts 1a and 1b). The elimination rate constant is the rate that the drug is removed from the body.
Time Frame: Day 28
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: 1/hour
Arm/Group | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid
Number analyzed (Participants) | 11 | 2
1/hour | 0.07 [0.06 to 0.09] | 0.09 [0.08 to 0.09]

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time of the baseline visit through Day 50.
Groups:
- Cohort 1a: Imatinib (50 mg): Participants in Cohort 1a while receiving 50 mg imatinib for 14 days.
- Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid: Participants in Cohort 1a while receiving 50 mg imatinib for 14 days together with rifabutin and isoniazid.
- Cohort 1b: Imatinib (100 mg): Participants in Cohort 1b while receiving 100 mg imatinib for 14 days.
- Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid: Participants in Cohort 1b while receiving 100 mg imatinib for 14 days together with rifabutin and isoniazid.
Arm/Group | Cohort 1a: Imatinib (50 mg) | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid | Cohort 1b: Imatinib (100 mg) | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid | Imatinib (100 mg)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14 | 0/6 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/6 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 16/16 | 12/14 | 5/6 | 3/3 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a: Imatinib (50 mg) (N=16) | Cohort 1a: Imatinib (50 mg) + Rifabutin + Isoniazid (N=14) | Cohort 1b: Imatinib (100 mg) (N=6) | Cohort 1b: Imatinib (100 mg) + Rifabutin + Isoniazid (N=3) | Imatinib (100 mg) (N=2)
Low Hemoglobin (Blood and lymphatic system disorders) | 9 | 1 | 1 | 1 | 1
Lymphopenia (low absolute lymphocyte count (ALC)) (Blood and lymphatic system disorders) | 2 | 4 | 1 | 3 | 1
Neutropenia (low absolute neutrophil count (ANC)) (Blood and lymphatic system disorders) | 0 | 1 | 0 | 3 | 1
White blood cell count decrease (Blood and lymphatic system disorders) | 2 | 5 | 0 | 2 | 0
Eosinophils increase (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Neutrophil decrease (Blood and lymphatic system disorders) | 6 | 3 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 2 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Edema localized (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 0
Elevated bilirubin (Hepatobiliary disorders) | 0 | 1 | 3 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 5 | 0 | 2 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 1
Hypoproteinemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 2 | 1 | 0 | 0 | 0
Menstrual disturbances (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0
Protein in urine (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urine discoloration (Renal and urinary disorders) | 0 | 4 | 0 | 0 | 0
Visual changes (General disorders) | 1 | 0 | 0 | 0 | 0
Bicarbonate low (General disorders) | 6 | 2 | 0 | 0 | 0
Blood urea nitrogen abnormal (General disorders) | 1 | 1 | 1 | 0 | 1
eGFR Decrease (General disorders) | 7 | 2 | 2 | 0 | 0
eGFR Decrease from Baseline (General disorders) | 3 | 1 | 0 | 0 | 0
Hypokalemia (General disorders) | 7 | 2 | 2 | 0 | 1
Hyponatremia (General disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Abdominal pain (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Headache (General disorders) | 1 | 0 | 0 | 1 | 0
Fever (General disorders) | 0 | 1 | 0 | 0 | 0
Mild heartburn (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Estimated creatinine clearance decrease from baseline (General disorders) | 0 | 0 | 0 | 0 | 1
Alkaline phosphatase (ALP) increase (General disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT03891901/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT03891901/ICF_001.pdf